CLINICAL TRIAL: NCT07360977
Title: A Composition Comprising Glucoraphanin, Myrosinase and a Buffered Solution for Use in the Treatment of Neurodegenerative Diseases
Brief Title: Myrosinase Bioactivated Gglucoraphanin for the Treatment of Neurodegenerative Diseases (GRA-MYR-ND)
Acronym: GRA-MYR-ND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Collaborators: Fondazione Edmund Mach (Other); Vittore Buzzi Children's Hospital (Other); Azienda Sanitaria Provinciale Ragusa (Other)
Responsible Party: Principal Investigator, Emanuela Mazzon, Professor, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GRA-MYR-ND; PNRR-POC-2022-12376049 (Other Grant/Funding Number: Funded by European Union-Next Generation EU-NRRP M6C2- investment 2.1)
Record Dates: First submitted 2025-12-18; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: PARKINSON DISEASE (Disorder); Multiple Sclerosis (MS) - Relapsing-remitting; Pediatric Patients Affected by Neuromuscolar and Degenerative Diseases
Keywords: phytocompounds; Glucosinolates; isothiocyanate; Parkinson's disease; multiple sclerosis
MeSH Terms: conditions — Parkinson Disease; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- PD patients receiving only standard therapy (No Intervention): Patients affected by Parkinson's disease receiving only standard therapy
- PD patients receiving bioactivated GRA (Experimental): Patients affected by Parkinson's disease receiving bioactivated GRA
  Interventions: Drug: bioactivated GRA for adult patients
- MS patients receiving only standard therapy (No Intervention): Patients affected by multiple sclerosis receiving only standard therapy
- MS patients receiving bioactivated GRA (Experimental): Patients affected by multiple sclerosis receiving bioactivated GRA
  Interventions: Drug: bioactivated GRA for adult patients
- Pediatric patients receiving only standard therapy (No Intervention): Pediatric patients receiving only standard therapy
- Pediatric patients receiving bioactivated GRA (Experimental): Pediatric patients receiving bioactivated GRA
  Interventions: Drug: bioactivated GRA for pediatric patients

INTERVENTIONS:
Drug: bioactivated GRA for adult patients — adult dose: 50 mg/day of bioactivated GRA for 6 months
  Arms: MS patients receiving bioactivated GRA; PD patients receiving bioactivated GRA
Drug: bioactivated GRA for pediatric patients — pediatric dose: 10 mg/day of bioactivated GRA for 6 months
  Arms: Pediatric patients receiving bioactivated GRA

SUMMARY:
Glucosinolates (GLs) are phytocompounds mainly found in the Cruciferae (Brassicacea) and Moringa oleifera plants. The hydrolysis of GLs by myrosinase led to the production of isothiocyanate (ITCs). ITCs consumption was associated with different health promoting effects, including to neuroprotective, anti-oxidant and anti-inflammatory capacities. In particular, they showed neuroprotective effects in experimental models of neurodegenerative diseases, including multiple sclerosis (MS) and Parkinson's disease (PD). From different GLs, different ITCs are originated. In particular, from glucoraphanin (GRA) the ITC sulforaphane (SFN) is obtained. The PI of the project is one of the proprietor of a patent (EP2908850B1) for the application of (Rs)-GRA with myrosinase in a buffered solution for the treatment of neurodegenerative diseases. The aim of this project is to evaluate the effects of the administration of bioactivated GRA in different cohorts of adult patients, affected by MS and PD, but also a cohort of pediatric patients affected by neuromuscolar and degenerative diseases. The effects of bioactivated (Rs)-GRA administration will be evaluated with a combination of clinical evaluations and a multiomic (metabolomic, genomic) approach.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for PD:

* Male or female patients aged between 45-75 years old.
* Clinical diagnosis of PD according to UK Brain Bank Criteria.
* 3 months of clinical stability before study enrolment.
* Anti-parkinsonian medication is fixed for at least 3 months prior to study entry.

Inclusion Criteria for MS:

* Male or female patients 18 years old or older.
* Diagnosis of RR-MS according to McDonald criteria.
* Expanded Disability Status Scale(EDSS) lower or equal to 5.5.
* Stable disease for at least 30 days prior to study entry.
* Stable disease-modifying therapy for at least 3 months prior to study entry.

Common inclusion criteria for MS and PD:

* No changes in drug treatment during 6 months-study treatment.
* Patients understand and comply with the study procedure and are able to complete tests and examinations required by the project.
* Written informed consent.

Inclusion criteria for pediatric patients:

* Eligible patients are those clinically stable;
* Age range from 1 to 10, between 5 and 30 kg.
* Patients not involved in other clinical trials.

Exclusion Criteria:

Exclusion criteria for PD and MS:

* Absolute contraindications to Magnetic Resonance Imaging (MRI).
* Concomitant neurological disease or severe co-morbidities able to influence outcomes such as spinal injury, cancer, dementia, or other central nervous system diseases such as stroke, epilepsy or psychiatric disorders;
* Total score of Mini-Mental State Examination (MMSE)<24.
* Participating in other clinical trials.
* Pregnant/lactating.

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-05-19 (Estimated); Study Completion 2026-05-19 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (UPDRS) Total Score | Baseline, 6 months (end of treatment), 12 months
  The score ranges from 0 to 260, with 0 indicating no disability and 260 indicating total disability. The scale is divided into four parameters: 0 (normal), 1 (mild), 2 (mild), 3 (moderate), and 4 (severe).
Hoehn and Yahr scale | Baseline, 6 months (end of treatment), 12 months
  Parkinson's Disease Progression Stage Scale (Stage 1 to 5). The scale is a subset of the Unified Parkinson's Disease Rating Scale, which allows for a more nuanced assessment of daily activities and non-motor symptoms in the context of disease therapy.
Expanded Disability Status Scale (EDSS) for Multiple Sclerosis patients | Baseline, 6 months (end of treatment), 12 months
  Evaluation of the degree of neurological disability in Multiple Sclerosis. The range of the EDSS Step includes 20 half steps from 0 to 10, with EDSS Step 0 corresponding to a completely normal examination and EDSS Step 10 to death due to MS
Cognitive and Neuropsychological Assessments: Montreal Cognitive Assessment (MoCA) and Mini-mental state examination | Baseline, 6 months (end of treatment), 12 months
  The MoCA is a one-page 30-point test administered in approximately 10 minutes to dectect cognitive impairment. Scores range between 0 and 30, a score of 26 or over is considered to be normal.
  The mini-mental state examination (MMSE) or Folstein test is a 30-point test to identify cognitive impairment. Any score of 24 or more (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment. The raw score may also need to be corrected for educational attainment and age
Brief Repeatable Battery (BRB) of Neuropsychological Tests for Multiple Sclerosis patients | Baseline, 6 months (end of treatment), 12 months
  THE BRB consists of twelve subtests which give five scores, one for each of the five domains tested (immediate memory, visuospatial/constructional, language, attention, delayed memory). Higher values represent a better outcome.
Normalized Brain Volume (NBV) | Baseline, 6 months (end of treatment), 12 months
  Evaluation of global brain atrophy through the measurement of total brain volume normalized for head size using high-field Magnetic Resonance Imaging (MRI). Higher values indicate better brain volume preservation, while a decrease over time indicates progression of brain atrophy.
Normalized Cortical Volume (NCV) | Baseline, 6 months (end of treatment), 12 months
  Evaluation of regional atrophy focusing on the cerebral cortex. Measurement of cortical gray matter volume normalized for head size using high-field MRI. This parameter is used to quantify the loss of cortical tissue specifically.
Change from Baseline in Whole-Brain Fractional Anisotropy (FA) in Multiple Sclerosis Patients | Baseline, 6 months (end of treatment), 12 months
  FA is a DTI-derived metric that reflects the microstructural integrity of white matter. In Multiple Sclerosis, a reduction in FA values is a marker of axonal damage and demyelination, even in Normal Appearing White Matter (NAWM).The unit of measurement is the Ratio (Scale from 0 to 1, where 1 indicates maximum diffusion/directional integrity.
Change from Baseline in Whole-Brain Mean Diffusivity (MD) in Multiple Sclerosis patients | Baseline, 6 months (end of treatment), 12 months
  MD measures the average magnitude of water diffusion. An increase in MD values in MS patients indicates loss of structural barriers, typically due to neurodegeneration, inflammation, or loss of myelin. This parameter provides a global index of tissue destruction.
Non-Motor Symptoms Scale (NMSS) for Parkinson patients | Baseline, 6 months (end of treatment), 12 months
  It assesses 30 non motor symptoms across 9 domains, with scores ranging from 0 (no symptoms) to 12 per group (severity x frequency), resulting in a total score of 0 to 360, indicating the extent of the non-motor symptom burden. Lower score indicate fewer symptoms; a negative change from baseline indicates improvement in symptoms. Mean scores vary with disease severity, reflecting increased problems with sleep disturbances, mood, cognition, gastrointestinal function, etc.
Quality of Life Assessment: Hamilton Rating Scale for Depression (HRSD) and Hamilton Anxiety Rating Scale. | Baseline, 6 months (end of treatment), 12 months
  Depression severity is assessed using the 17-item Hamilton Rating Scale for Depression (HRSD). Based on the total score, participants will be classified into the following levels: no depression (0-7), mild depression (8-13), moderate depression (14-18), severe depression (19-22), and very severe depression (≥23). The Hamilton Anxiety Rating Scale (HAM-A) is a psychological questionnaire to evaluate the anxiety. The Hamilton Anxiety Rating Scale (HAM-A), which consists of 14 items, each rated on a 5-point scale. The total score, obtained by adding the individual items, ranges from 0 to 56. A score ≤17 indicates mild anxiety; 18-24 indicates mild to moderate anxiety; 25-30 indicates moderate to severe anxiety.
Parkinson's Disease Quality of Life Questionnaire (PDQ-8) | Baseline, 6 months (end of treatment), 12 months
  It is a patient-reported outcome measure consisting of 8 items that assesses health-related quality of life in Parkinson's disease. It includes one representative item for each domain of the original PDQ-39: mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication, and physical discomfort. Participants rate their experiences in the previous month using a 5-point Likert scale (0 = never to 4 = always). The total score is converted into a Summary Index (SI) ranging from 0 to 100, with higher scores indicating poorer health-related quality of life.Summary Index scores were interpreted as follows: 0-20 indicating good quality of life with minimal disease impact, 21-40 mild impairment, 41-60 moderate impairment, 61-80 marked impairment, and 81-100 severe impairment of quality of life.
Parkinson's Disease Sleep Scale (PDSS-2) | Baseline, 6 months (end of treatment), 12 months
  The PDSS-2 is a 15-item self-administered questionnaire used to evaluate sleep disturbances and nocturnal symptoms in patients with Parkinson's Disease. It covers various domains including motor symptoms at night, sleep quality, and daytime sleepiness. Each item is scored on a 5-point Likert scale from 0 (never) to 4 (very often). The total score ranges from 0 to 60. A total score ≥ 15-18 is often considered indicative of clinically significant sleep disturbance.
Change from Baseline in EuroQol-5D-3L Index Score | Baseline, 6 months (end of treatment), 12 months
  The EQ-5D-3L is a standardized instrument for measuring health-related quality of life. It consists of a questionnaire with 5 item: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. These responses are converted into a single index score (utility value) using a country-specific value set.
Clinical Global Impression of Improvement (CGI-I) | Baseline, 6 months (end of treatment), 12 months
  The CGI-I is a clinician-rated scale that assesses how much the patient's illness has improved or worsened relative to a baseline state.It is scored on a 7-point Likert scale: 1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no change from baseline (the initiation of treatment); 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment
Patient Global Impression of Change (PGI-C) | Baseline, 6 months (end of treatment), 12 months
  The PGI-C is a self-reported scale reflecting the patient's belief about the efficacy of treatment and their overall change in health status since the start of the study. It uses a 7-point scale where: 1 = Very much improved; 2 = Much improved; 3 = Minimally improved; 4 = No change; 5 = Minimally worse; 6 = Much worse; 7 = Very much worse.

SECONDARY OUTCOMES:
Changes in growth parameters, anthropometric measurements and pubertal status. | Baseline, 3 , 6 (end of the treatment) , and 12 months
  Evaluation of physical development and nutritional status. The following parameters will be measured: body weight (kg), height (cm), Body Mass Index (BMI, calculated as weight in kilograms divided by height in meters squared), and their respective percentiles adjusted for age, sex, and specific pathology. These measurements aim to assess the impact of the administration of the study composition on growth and development in the pediatric population. Additionally, pubertal development will be assessed using the Tanner Stage (Sexual Maturity Rating), which evaluates the progression of secondary sexual characteristics (breast development in girls, genital development in boys, and pubic hair in both) on a scale from 1 (pre-pubertal) to 5 (adult). This combined assessment aims to monitor the global growth trajectory and hormonal-physical maturation during the treatment.
Changes in Electroencephalogram (EEG) Mean Frequency and Brain Electrical Activity. | Baseline, 3, 6 ( end of the treatment), 12 months
  Evaluation of cerebral electrical activity using the Micromed Brain Quick System (System Plus Evolution software) with a 48-channel recording head. Recordings will follow the International 10-20 system (or reduced electrode sets for infants < 40 cm). The signal will be processed with a sampling frequency of 256 Hz, a high-pass filter of 1.6 Hz, a low-pass filter of 30 Hz, and a sensitivity of 100 μV/cm. Assessments will include wakefulness, sleep deprivation, and afternoon rest. For patients with severe neurological conditions, video-EEG and polygraphy will be associated. The analysis focuses on background activity evolution and paroxysmal abnormalities according to ILAE guidelines.Unit of Measure: Qualitative and Quantitative neurophysiological parameters (presence/absence of epileptiform activity and mean frequency in Hz.
Assessment of Swallowing Function via Dysphagia Outcome and Severity Scale (DOSS) in pediatric patients. | baseline and 3, 6, 12 months
  Evaluation of the severity of dysphagia (swallowing impairment). The DOSS is a 7-point scale used to systematically rate functional longitudinal changes in swallowing. Scores range from 1 (Severe dysphagia: nothing by mouth) to 7 (Normal in all situations).
Changes in Psychomotor Development via Griffiths Mental Development Scales 3 (GMDS-3) | baseline and 3, 6, 12 months.
  The Griffiths-3 Scale (Griffiths III) is a comprehensive developmental assessment for young children (birth to nearly 6 years) that measures mental and physical growth across five key domains: Foundations of Learning, Language & Communication, Eye & Hand Coordination, Personal-Social-Emotional, and Gross Motor.Unit of Measure: Developmental Quotient (DQ) score (Standardized score where the mean is 100 and the standard deviation is 15. Higher scores indicate more advanced development).
Pediatric Esophageal Motility and Dysphagia Assessment via High-Resolution Manometry (HRM). | baseline and 3, 6 ( end of the treatment), 12 months
  Evaluation of oro-pharyngeal and esophageal motility using the HRM ManoScan™ ESO System. The procedure uses a catheter (max diameter 2.75 mm to 4.2 mm, selected based on age/weight) and follows international standards (e.g., German Guidelines for neurogenic dysphagia). Key metrics include the characterization of esophageal function and the study of the esophagogastric junction motility.Unit of Measure: Composite Score and Manometric Parameters (including mmHg for pressures and Chicago Classification v4.0 metrics).
Metabolomics and Pharmacokinetic Analysis of Bioactive Compounds and Endogenous Metabolites in pediatric, PD and MS patients | baseline and 6 months (end of treatment)
  Evaluation of the metabolic profile in human biofluids (plasma and urine) using Liquid Chromatography-Mass Spectrometry (LC-MS). The analysis includes:
  Exogenous Compound Tracking: Determination of the metabolic fate and bioavailability of the administered phytocompound (Glucoraphanin/Sulforaphane).
  Targeted Plasma Metabolomics: Quantitative analysis of essential amino acids (Tryptophan, Tyrosine, Phenylalanine) and their catabolites.
  Microbiota-Derived Metabolites: Assessment of Short-Chain Fatty Acids (SCFAs) and Medium-Chain Fatty Acids (MCFAs) in plasma as indicators of gut microbiota modulation.
  Urinary Endogenous Metabolites: Evaluation of changes in the urinary metabolic fingerprint to identify biomarkers of response to treatment.
Transcriptomic Profile and Differential Gene Expression Analysis for PD,MS and pediatric patients. | baseline and 6 months (end of treatment)
  Evaluation of gene expression changes in response to the study treatment. RNA sequencing (RNA-seq) will be performed using Illumina platforms. The bioinformatics pipeline includes:Data Quality Control: FastQC for raw data assessment. Preprocessing: Trimmomatic for adapter trimming and quality filtering.Alignment: STAR aligner against the GRCh38 human reference genome.
  Quantification: Transcript counting via the HTSeq-count package. Differential Expression: Identification of Differentially Expressed Genes (DEGs) using the DESeq2 library in R. Statistical analysis: To ensure robustness, false positives will be controlled using the Benjamini-Hochberg post-hoc procedure with a significance threshold (q-value) set at 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Emanuela Mazzon, Principal Investigator — IRCCS Centro Neurolesi Bonino Pulejo
Locations (1):
- IRCCS Centro Neurolesi Bonino Pulejo, Messina, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deuschl G, Beghi E, Fazekas F, Varga T, Christoforidi KA, Sipido E, Bassetti CL, Vos T, Feigin VL. The burden of neurological diseases in Europe: an analysis for the Global Burden of Disease Study 2017. Lancet Public Health. 2020 Oct;5(10):e551-e567. doi: 10.1016/S2468-2667(20)30190-0. PMID 33007212
- [Background] Klomparens EA, Ding Y. The neuroprotective mechanisms and effects of sulforaphane. Brain Circ. 2019 Apr-Jun;5(2):74-83. doi: 10.4103/bc.bc_7_19. Epub 2019 Jun 27. PMID 31334360
- [Background] Yadav SK, Soin D, Ito K, Dhib-Jalbut S. Insight into the mechanism of action of dimethyl fumarate in multiple sclerosis. J Mol Med (Berl). 2019 Apr;97(4):463-472. doi: 10.1007/s00109-019-01761-5. Epub 2019 Feb 28. PMID 30820593
- [Background] Kamal RM, Abdull Razis AF, Mohd Sukri NS, Perimal EK, Ahmad H, Patrick R, Djedaini-Pilard F, Mazzon E, Rigaud S. Beneficial Health Effects of Glucosinolates-Derived Isothiocyanates on Cardiovascular and Neurodegenerative Diseases. Molecules. 2022 Jan 19;27(3):624. doi: 10.3390/molecules27030624. PMID 35163897
- [Background] Schepici G, Bramanti P, Mazzon E. Efficacy of Sulforaphane in Neurodegenerative Diseases. Int J Mol Sci. 2020 Nov 16;21(22):8637. doi: 10.3390/ijms21228637. PMID 33207780
- [Background] Lotti C, Rubert J, Fava F, Tuohy K, Mattivi F, Vrhovsek U. Development of a fast and cost-effective gas chromatography-mass spectrometry method for the quantification of short-chain and medium-chain fatty acids in human biofluids. Anal Bioanal Chem. 2017 Sep;409(23):5555-5567. doi: 10.1007/s00216-017-0493-5. Epub 2017 Jul 17. PMID 28717897
- [Background] Garcia-Aloy M, Ulaszewska M, Franceschi P, Estruel-Amades S, Weinert CH, Tor-Roca A, Urpi-Sarda M, Mattivi F, Andres-Lacueva C. Discovery of Intake Biomarkers of Lentils, Chickpeas, and White Beans by Untargeted LC-MS Metabolomics in Serum and Urine. Mol Nutr Food Res. 2020 Jul;64(13):e1901137. doi: 10.1002/mnfr.201901137. Epub 2020 Jun 22. PMID 32420683
- [Background] Ulaszewska, M.M., Trost, K., Stanstrup, J. et al. Urinary metabolomic profiling to identify biomarkers of a flavonoid-rich and flavonoid-poor fruits and vegetables diet in adults: the FLAVURS trial
- [Background] Anesi A, Berding K, Clarke G, Stanton C, Cryan JF, Caplice N, Ross RP, Doolan A, Vrhovsek U, Mattivi F. Metabolomic Workflow for the Accurate and High-Throughput Exploration of the Pathways of Tryptophan, Tyrosine, Phenylalanine, and Branched-Chain Amino Acids in Human Biofluids. J Proteome Res. 2022 May 6;21(5):1262-1275. doi: 10.1021/acs.jproteome.1c00946. Epub 2022 Apr 5. PMID 35380444